CLINICAL TRIAL: NCT01647971
Title: An Open Label Phase I/II Study of the Efficacy and Safety of Ublituximab in Patients With B-cell Non-Hodgkin Lymphoma Who Have Relapsed or Are Refractory After CD20 Directed Antibody Therapy
Brief Title: Study of the Efficacy and Safety of Ublituximab in Patients With Relapsed or Refractory B-cell Non-Hodgkin Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: TG Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TGTX 1101-101
Record Dates: First submitted 2012-07-17; First posted 2012-07-24 (Estimated); Last update posted 2022-11-21 (Actual); Status verified 2022-11

CONDITIONS: Non-Hodgkins Lymphoma; B-cell Lymphoma; Waldenstrom's Macroglobulinemia; Marginal Zone Lymphoma; Chronic Lymphocytic Leukemia (CLL); Small Lymphocytic Lymphoma (SLL); Primary Central Nervous System Lymphoma
Keywords: Lymphoma; Rituxan; Relapsed; Refractory
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, B-Cell; Waldenstrom Macroglobulinemia; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma; Recurrence | interventions — ublituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ublituximab (Experimental): Phase I:
  4 cohorts with IV ublituximab starting with 450 mg followed by 600 mg, 900 mg or 1200 mg in each cohort (3 - 6 patients per cohort). Infusions will be on days 1, 8, 15 and 22 of cycle 1 followed by a planned maintenance with a single infusion monthly starting cycle 3. Patients with chronic lymphocytic leukemia (CLL) or small lymphocytic lymphoma (SLL) will have infusions on Days 1, 8 and 15 of cycle 1 & 2 followed by a planned maintenance with a single infusion monthly starting cycle 3. Expansion of patient enrollment in select cohorts will apply.
  Interventions: Drug: Ublituximab

INTERVENTIONS:
Drug: Ublituximab — Ublituximab is a novel monoclonal antibody targeting cluster of differentiate 20 (CD20)

SUMMARY:
The purpose of this study is to determine whether ublituximab is safe and effective in patients with relapsed or refractory B-cell lymphoma who were previously treated with rituximab.

ELIGIBILITY:
Inclusion Criteria:

* Relapsed or Refractory B-cell Lymphoma
* Measurable or Evaluable Disease
* Previously treated with at least one line of rituximab or a rituximab based therapy
* Patients ineligible for high dose or combination chemotherapy + stem cell transplant
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0, 1 or 2
* No active or chronic infection of Hepatitis B or C and no history of HIV based on negative serology

Exclusion Criteria:

* Prior chemotherapy, investigational therapy or radiotherapy within 3 weeks of study entry
* Prior autologous or allogeneic stem cell transplantation within 3 months of study entry
* History of severe hypersensitivity or anaphylaxis to prior rituximab
* Uncontrolled inter-current illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, brain metastasis, or psychiatric illness that would limit compliance with study requirements
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2012-07-19 (Actual); Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | Subjects will be followed for 4 weeks
  Safety for all study patients will be evaluated by a Data Safety Monitoring Board to determine if feasible to continue with dose escalation
Maximum Tolerated Dose acceptable for participants | Subjects will be followed for 4 weeks
  The Maximum Tolerated Dose will be determined by a Data Safety Monitoring Board

SECONDARY OUTCOMES:
Efficacy | Participants will be evaluated approximately every 8 - 12 weeks
  Efficacy will include overall response rate, duration of response and progression-free survival

OTHER OUTCOMES:
Pharmacokinetic profile including Peak Plasma Concentration (Cmax)" or "Area Pharmacokinetic profile including Peak Plasma Concentration (Cmax) and Area under the plasma concentration versus time curve (AUC) | Up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: TG Therapeutics Clinical Trials, Study Director — TG Therapeutics, Inc.
Locations (8):
- United States (8):
  - TG Therapeutics Investigational Trial Site, Huntsville, Alabama
  - TG Therapeutics Investigational Trial Site, Jonesboro, Arkansas
  - TG Therapeutics Investigational Trial Site, Athens, Georgia
  - TG Therapeutics Investigational Trial Site, Macon, Georgia
  - TG Therapeutics Investigational Trial Site, Bethesda, Maryland
  - TG Therapeutics Investigational Trial Site, Morristown, New Jersey
  - TG Therapeutics Investigational Trial Site, New York, New York
  - TG Therapeutics Investigational Trial Site, Memphis, Tennessee